CLINICAL TRIAL: NCT06799273
Title: MECKI-Amyloidosis: Assessment of the Exercise Capacity and Prognosis of Patients with Cardiac Amyloidosis
Acronym: MECKI-AMI
Status: Recruiting | Type: Observational
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Sponsor
Other Study IDs: MECKI-AMYLOIDOSIS
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Amyloidosis patients (prospective cohort): Prospectively enrolled patients diagnosed with cardiac amyloidosis
- Heart Failure patients (retrospective cohort): Patients with history of heart failure with reduced ejection fraction previously enrolled in the MECKI score registry

SUMMARY:
This study aims to advance the understanding of cardiac amyloidosis, its effects on exercise capacity, and its prognostic implications. By conducting a systematic investigation with particular emphasis on longitudinal evaluation, we aim to provide valuable insights to guide clinical practice and improve the management of patients with cardiac amyloidosis.

Our study intends to follow patients for a period of two years, evaluating them every six months. This longitudinal approach allows us to monitor changes in exercise capacity and other relevant clinical parameters over time. Furthermore, it enables the development of a prognostic tool similar to the MECKI score, capable of assessing the risk of adverse events in patients with cardiac amyloidosis based on their exercise performance.

By comparing our results with data from heart failure patients already included in the MECKI score database, we also aim to highlight any differences in prognosis between patients with cardiac amyloidosis and those with general heart failure. Finally, we aim to characterize cardiac amyloidosis by differentiating it from general heart failure. By comparing our results with data from heart failure patients already included in the MECKI score database, we can clarify the distinct exercise limitations in cardiac amyloidosis and shed light on how they differ from more conventional heart failure.

ELIGIBILITY:
Inclusion criteria

* Age > 18 years
* Diagnosis of cardiac amyloidosis obtained by MRI or scintigraphy
* Ability to perform a cardiopulmonary exercise test

Exclusion criteria

* severe obstructive pulmonary disease
* exercise-induced angina
* significant ECG changes
* presence of clinical comorbidities that interfere with exercise performance

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective Cohort: Patients with Diagnosis of cardiac amyloidosis.
  Retrospective cohort:
  Population of heart failure patients selected from the MECKI score database
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the parameters most closely correlated with two-year prognosis in patients with cardiac amyloidosis in order to create a specific risk score for these patients. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Cardiologico Monzino, Irccs, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No